CLINICAL TRIAL: NCT06234553
Title: Radiomics-based Diagnosis, Treatment and Outcome Prediction for Pituitary Adenoma
Brief Title: Application of Radiomics in the Diagnosis and Treatment Prediction of Pituitary Adenoma
Acronym: RIPA
Status: Active, not recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SK-748; RIPA-001 (Other: tiantan hospital)
Record Dates: First submitted 2023-12-18; First posted 2024-01-31 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- training set and validation set: Retrospective study focusing on the diagnosis and treatment outcomes of pituitary adenomas
  Interventions: Procedure: surgery of pituitary adenomas

INTERVENTIONS:
Procedure: surgery of pituitary adenomas — evaluate pathological type and treatment effect after treatment

SUMMARY:
The images of patients with Pituitary adenoma were collected and analyzed based on the methods of radiomics.

DETAILED DESCRIPTION:
Inclusion of pituitary adenoma patients diagnosed clinically or pathologically

1. Clinical data and pre-treatment imaging data of included patients (DICOM format)
2. Determine the subtype diagnosis of pituitary adenoma based on the patient's clinical and pathological data
3. Collect relevant data of patients before and after treatment
4. Using radiomics methods, extract radiomic features of patients and construct a radiomic model for predicting the diagnosis and treatment response of pituitary adenomas

ELIGIBILITY:
Inclusion Criteria:

1. Gender unlimited, 18-80 years old;
2. Clinical diagnosis of Pituitary Adenoma and receive surgical treatment;
3. Received brain imaging;
4. informed consent signed

Exclusion Criteria:

1. Pregnant / lactating women
2. Contraindications of imaging examination
3. Lack of effective clinical data
4. MRI data before treatment cannot be obtained
5. Postoperative pathology not revealed pituitary adenoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants willing to receive brain imaging could be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate of pituitary adenoma | 1 year after treatment
  The pituitary adenoma recurred 1 year after treatment. The recurrence was assessed by 3 aspects: (1)contrast enhanced MRI showed suspicious tumor growth, such as bone destruction; (2)signs and symptoms that had disappeared after treatment reappeared, such as pressing on nearby nerve tissue and some characteristic appearance; (3)endocrine indexes rose again after reaching the remission standard, iculding Prolactin(PRL)>30 μg/L in Lactotroph adenoma; growth hormone (GH)>2.5ng/ml in Somatotroph adenoma, serum cortisol>800nmol/L at 8am in Corticotroph adenoma, while other types do not consider endocrine indicators.

SECONDARY OUTCOMES:
Pathological type of pituitary adenomas | 1 week after treatment
  The pathological examination was used to evaluated the type of pituitary adenoma. The pathological type was assessed by 2017 WHO standard, divided into Somatotroph adenoma, Lactotroph adenoma, Thyrotroph adenoma, Corticotroph adenoma, Gonadotroph adenoma, Null-cell adenoma and Plurihormonal and double adenomas.

CONTACTS AND LOCATIONS:
Overall Officials: Yanghua Fan, Dr., Study Director — Beijing Tiantan Hospital
Locations (1):
- Beijing tiantan hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No